CLINICAL TRIAL: NCT06075641
Title: Comparison of Surgical Stripping and Erbium, Chromium:Yttrium-scandium-gallium-garnet (Er,Cr:YSGG) Laser Techniques for Gingival Depigmentation Recurrence: A Randomized Clinical Trial, Four Years Follow up
Brief Title: Post Gingival Depigmentation Assessment: Comparison of Surgical Stripping vs (Er,Cr:YSGG) Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Talal Zahid, Chairman of Periodontology Department, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 077-16
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Pigmentation; Gingiva
Keywords: gingival pigmentation; depigmentation; Er,Cr:YSGG; laser
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical Stripping (Active Comparator)
  Interventions: Procedure: Gingival depigmentation
- Erbium, chromium:yttrium-scandium-gallium-garnet (Er,Cr:YSGG) Laser Techniques (Experimental)
  Interventions: Procedure: Gingival depigmentation

INTERVENTIONS:
Procedure: Gingival depigmentation — Gingival depigmentation is the most widely used periodontal procedure to remove or reduce the melanotic areas. Various techniques can be employed to effectively carry out the depigmentation procedure, including surgical scraping, scalpel technique, bur abrasion, free gingival graft, gingivectomy, cryosurgery, electrosurgery, chemical therapies, and different types of lasers

SUMMARY:
The appearance and health of the gingiva significantly contribute to an aesthetically pleasing smile. Pink gingiva indicates healthy gums and is generally preferred over dark or mixed colors. However, gingival color varies among individuals based on factors such as race, geography, gum health, epithelial thickness, vascular supply, keratinization level, and pigments in the epithelium layers.

Four primary pigments define mucosa color: melanin, oxygenated hemoglobin (Hb), carotenoids, and reduced Hb. Melanin notably affects excessive gingival pigmentation. Gingival melanin hyperpigmentation, sometimes called racial pigmentation, is a genetic trait present in many ethnic groups due to excess melanin deposition in the epithelial layers. While not a medical concern, this hyperpigmentation can be unattractive, especially for those with a gummy smile. As a result, many seek treatments to reduce or eliminate this pigmentation.

Various methods for gingival depigmentation exist, including surgical scraping, scalpel technique, bur abrasion, free gingival graft, gingivectomy, cryosurgery, electrosurgery, chemical treatments, and lasers. A significant challenge with these treatments is gingival repigmentation or the reappearance of melanin post-procedure.

For years, the scalpel technique was the standard. It's a straightforward and economical method that involves removing the gingival epithelium and some underlying tissue. Although it promotes quick healing, the procedure can cause bleeding, necessitating local anesthesia and post-operative dressings. Due to the associated discomfort, researchers have sought equally effective alternatives.

Laser ablation has become a popular choice among dental professionals and patients. Lasers like carbon dioxide (CO2), diode, argon, ruby, Nd:YAG (neodymium-doped yttrium aluminum garnet) , and Er:YAG (erbium-doped yttrium aluminium garnet) have been proven effective through numerous studies. Lasers present benefits such as minimal post-operative pain, ease of use, and quicker treatment times. Recurrence rates post-laser surgery (1.16%) are lower than with the scalpel technique (4.25%). However, lasers also have downsides, including high costs, potential for thermal damage, and the risk of deep penetration.

One laser, the Erbium-chromium:yttrium-scandium-gallium-garnet (Er,Cr:YSGG), has been FDA-approved for certain dental procedures but hasn't been widely used for gingival depigmentation. Preliminary findings suggest it offers advantages like reduced pain and faster healing compared to other lasers. In a case study involving two patients, the Er,Cr:YSGG laser effectively removed gingival pigmentation, with no recurrence observed after six months.

This clinical trial aimed to compare the efficacy and recurrence rates between the conventional scalpel technique and the Er,Cr:YSGG laser technique. The hypothesis suggests that the Er,Cr:YSGG laser might be a superior treatment for gingival hyperpigmentation compared to other methods.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Periodontally healthy subjects with concerns about their esthetics and presence of gingival hyperpigmentation in the upper arch

Exclusion Criteria:

* (1) smokers or were previous smokers
* (2) had a systemic disease/condition,
* (3) were pregnant/lactating
* (4) had gingivitis, periodontitis or any other periodontal disease
* (5) acquired amalgam pigmentation were excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Oral pigmentation index (DOPI) | Pre surgical, 1 month post op, 12 months post op
  This index of oral pigmentation is the commonly used index due to its simplicity and ease of use. The scores are as follows:
  0 = No clinical pigmentation (pink-colored gingiva)
  1. Mild clinical pigmentation (mild light brown color)
  2. Moderate clinical pigmentation (medium brown or mixed pink and brown color)
  3. Heavy clinical pigmentation (deep brown or bluish black color)
Gingival melanosis record (GMR) | Pre surgical, 1 month post op, 12 months post op
  A quantitative analysis method using clinical oral photographs